CLINICAL TRIAL: NCT04038710
Title: An Observational Study of the Effects on Clinical Outcomes of Expanded Access Program of Vertex Triple Combination Therapy.
Brief Title: Clinical Outcomes of Triple Combination Therapy in Severe Cystic Fibrosis Disease.
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: HS-3235
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with severe disease: Patients that are eligible to enroll in Vertex's triple combination therapy through the expanded access program.
  Interventions: Drug: Triple combination therapy

INTERVENTIONS:
Drug: Triple combination therapy — Triple combination is compromised of the drugs ivacaftor, tezacaftor and Vertex's next generation modulator.

SUMMARY:
This is an observational study of people with severe cystic fibrosis that are eligible for Vertex's triple combination therapy through its expanded access. Pulmonary health, intestinal health, and the overall health of individuals will be tracked for a year to see how effective triple combination therapy is in these people with severe cystic fibrosis disease.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Cystic Fibrosis
* Ability to reproducibly perform spirometry (according to ATS criteria)
* Physician decision to treat with TCT through the EAP program
* Ability to understand and sign a written informed consent or assent and comply with the requirements of the study

Exclusion Criteria:

* History of hypersensitivity to VX 445, VX 659, tezacaftor and/or ivacaftor
* Any acute lower respiratory symptoms treated with oral, inhaled or IV antibiotics or systemic corticosteroids within the 2 weeks prior to Visit 1.
* Major or traumatic surgery within 12 weeks prior to Visit 1.
* Initiation of any new chronic therapy (e.g., ibuprofen, Pulmozyme®, hypertonic saline, azithromycin, TOBI®, Cayston®) within 4 weeks prior to Visit 1.
* Use of an investigational agent within 28 days prior to Visit 1.
* History of lung or liver transplantation or listing for organ transplantation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at National Jewish Health with Cystic Fibrosis who are eligible to enroll in Vertex's triple combination therapy expanded access program.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
pulmonary function | For a year post initiation of therapy.
  FEV1 values.

SECONDARY OUTCOMES:
CFQ-R score | For a year following the initiation of triple combination therapy.
  cystic fibrosis questionnaire - revised has sections to measure pulmonary health and gastrointestinal health.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Low, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No